CLINICAL TRIAL: NCT01265043
Title: A Randomized Clinical Trial of Oral Health Promotion Interventions Among Patients Following Stroke
Brief Title: A Randomized Clinical Trial of Oral Health Promotion Interventions Among Patients After Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Otto Lok-Tao Lam, Clinical assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKCTR-1159
Record Dates: First submitted 2010-12-07; First posted 2010-12-22 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Acute Stroke
Keywords: oral health; oral hygiene; bacteria; quality of life; Clinical oral health in patients following acute stroke; Oral opportunistic pathogens in patients following acute stroke; Oral health-related quality of life in patients following acute stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OHI (Experimental): Patients provided with oral hygiene instruction and electric toothbrush
  Interventions: Other: Oral hygiene intervention
- OHI + CHX mouthrinse (Experimental): Patients provided with oral hygiene instruction and Corsodyl mouthrinse
  Interventions: Other: Oral hygiene intervention
- OHI + CHX mouthrinse + assisted brushing (Experimental): Oral hygiene instruction, Corsodyl mouthrinse, and assisted brushing
  Interventions: Other: Oral hygiene intervention

INTERVENTIONS:
Other: Oral hygiene intervention — Oral health promotion intervention

SUMMARY:
The main aim of this oral health intervention project is to compare the effect of providing 1) professional oral hygiene instruction alone versus 2) professional oral hygiene instruction plus adjunctive Chlorhexidine mouth rinse versus 3) professional oral hygiene instruction plus adjunctive assisted tooth brushing and Chlorhexidine mouth rinse, on the oral health condition, the general health condition and health-related quality of life (HRQoL) of patients with stroke who are receiving hospital-based rehabilitation. An additional aim is to assess potential longer term oral intervention-related health and HRQoL outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and over
* Moderate to severe stroke (Barthel Index >/= 70)
* Admitted to Rehabilitation Unit within 7 days

Exclusion Criteria:

* Patients with naso-gastric feeding tube
* Edentulous patients
* Patients with communication difficulties

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in plaque scores over course of trial | Three week in-hospital rehabilitation period

SECONDARY OUTCOMES:
Change in gingival bleeding scores over course of trial | three week in-hospital rehabilitation period
Change in oral colonization by aerobic and facultatively anaerobic Gram-negative bacilli over course of trial | Three week in-hospital rehabilitation period
Change in oral colonization by Staphylococcus aureus over course of trial | Three week in-hospital rehabilitation period
Change in oral colonization by yeasts over course of trial | Three week in-hospital rehabilitation period
Change in health-related quality of life over course of trial | three week in-hospital rehabilitation period
Change in oral health-related quality of life over course of trial | Three week in-hospital rehabilitation period

CONTACTS AND LOCATIONS:
Overall Officials: Otto LT Lam, BDS, BSc, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Tung Wah Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lam OL, McMillan AS, Samaranayake LP, Li LS, McGrath C. Effect of oral hygiene interventions on opportunistic pathogens in patients after stroke. Am J Infect Control. 2013 Feb;41(2):149-54. doi: 10.1016/j.ajic.2012.02.020. Epub 2012 Jul 17. PMID 22818804